CLINICAL TRIAL: NCT04542746
Title: The Role of Surgical Flap Design on the Healing of Intraosseous Defects Treated by Means Regenerative Therapy. Randomized Controlled Clinical Trial.
Brief Title: Treatment of Periodontal Intraosseous Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iorio Research and Dental Practice (Other)
Responsible Party: Principal Investigator, Vincenzo Iorio-Siciliano, DDS,PhD, Iorio Research and Dental Practice
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0012240
Record Dates: First submitted 2020-07-30; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive surgical technique (Experimental): The intra-bony defects of subjects allocated in test group were treated with a combination of minimally invasive surgical technique (MIST) and enamel matrix derivative( EMD).
  Interventions: Procedure: Minimally invasive surgical technique
- Conventional open flap debridement with papilla preservation (Active Comparator): The intra-bony defects of control group were treated using a combination of conventional open flap debridement with papilla preservation (COFD+PP) and EMD.
  Interventions: Procedure: Minimally invasive surgical technique

INTERVENTIONS:
Procedure: Minimally invasive surgical technique — After local anesthesia , for the sites of test group , a minimally invasive surgical technique (MIST) will be performed. The defects associated inter-dental papilla will be surgically approached with a diagonal incision following the pattern of the simplified papilla preservation flap. Flap elevation was to the buccal and oral aspect in the interdental space, An enamel matrix derivative (EMD) was applied into the defect.f A primary closure of the interdental papillae will be achieved using a 5-0 monofilament non resorbable suturing material.
  Other Names: Conventional open flap debridement with papilla preservation

SUMMARY:
The aim of the present study was to evaluate the impact of surgical flap design on the healing of intrabony defects treated by means periodontal regeneration. Forty patients were enrolled and allocated random in two groups. Patients of test group received a minimally invasive surgical flap , while patients of control group received a conventional access flap. In both group the intrabony were treated by means the same periodontal regeneration procedure (i.e application of enamel matrix derivative). Periodontal parameters were recoded at baseline and after 12-months observation time.

DETAILED DESCRIPTION:
This study was designed as multicenter randomized control clinical trial. The present trial was conduced according to CONSORT statement for improving the quality of reports of parallel-group randomized trials .

The intra-bony defects of subjects allocated in test group were treated with a combination of minimally invasive surgical technique (MIST) and enamel matrix derivative(EMD), while the intra-bony defects of control group were treated using a combination of conventional open flap debridement with papilla preservation (COFD+PP) and EMD.

Primary outcome

The primary outcome was based on Clinical attachment level gain( CAL gain)

Null hypothesis

Statistically significant different in terms of CAL gain will be recorded between test and control procedures.

Sample Size Calculation

The investigators are planning a study of a continuous response variable from independent control and experimental subjects with 1 control per experimental subject. In a previous study the response within each subject group was normally distributed with standard deviation 0,92. If the true difference in the experimental and control means is 0,97, we will need to study 20 experimental subjects and 20 control subjects to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0,8. The Type I error probability associated with this test of this null hypothesis is 0,05. Twenty-six patients were enrolled in the study and allocated in test or control group. In each patients 1 intra-bony defect was considered.

Randomization

The patients were randomly assigned to one of the two experimental procedures. The allocation was carried out using a commercially available computer software package. Treatment allocation was performed at time of surgery by opening an envelope containing the information test (i.e.EMD + MIST) or control (i.e.EMD + COFD+PP) procedure, respectively.

Inclusion Criteria

* Patients suffering from chronic periodontitis;
* Male and female ;
* Age 18 years old;
* Presence of intra-bony defects (contained and non-contained defects) in either the maxilla or the mandible with a PD ≥ 6 mm.
* II and III wall Intra-bony defects with an intra-bony component range from 3 mm to 6 mm for both groups;
* Intra-bony defect located only at one aspect ( mesial or distal)

Exclusion Criteria

* Patients with systemic disease;
* Prolonged antibiotic treatment or anti-inflammatory treatment within 4 weeks prior to surgery;
* Pregnant or lactating;
* Tobacco smokers;
* Patients with FMPS and FMBS 25 % after completion of non surgical periodontal therapy (recorded at six sites per tooth);
* Furcations;
* Third molars
* Teeth with circumferencial defects
* I-wall intra-bony defects

ELIGIBILITY:
Inclusion Criteria:

* • Patients suffering from chronic periodontitis;

  * Male and female ;
  * Age 18 years old;
  * Presence of intra-bony defects (contained and non-contained defects) in either the maxilla or the mandible with a PD ≥ 6 mm.
  * II and III wall Intra-bony defects with an intra-bony component range from 3 mm to 6 mm for both groups;
  * Intra-bony defect located only at one aspect ( mesial or distal)

Exclusion Criteria:

* • Patients with systemic disease;

  * Prolonged antibiotic treatment or anti-inflammatory treatment within 4 weeks prior to surgery;
  * Pregnant or lactating;
  * Tobacco smokers;
  * Patients with FMPS and FMBS 25 % after completion of non surgical periodontal therapy (recorded at six sites per tooth);
  * Furcations;
  * Third molars
  * Teeth with circumferencial defects
  * I-wall intra-bony defects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-08-12 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level gain ( CAL gain) | At 12 months
  Vertical measure from the cement enamel junction to the bottom of the defect.

CONTACTS AND LOCATIONS:
Locations (1):
- Iorio Research and Dental Practice, Naples, Italy